CLINICAL TRIAL: NCT05178186
Title: Impact of the COVID-19 Pandemic on Surgery for Thyroid Cancer: an International Multicenter Study
Brief Title: Impact of the COVID-19 Pandemic on Surgery for Thyroid Cancer
Acronym: THYCOVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Fabio Medas, Associate Professor, University of Cagliari
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: THYCOVID
Record Dates: First submitted 2021-12-30; First posted 2022-01-05 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Thyroid Carcinoma
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Thyroidectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Thyroid carcinoma (Other): Patients with thyroid carcinoma submitted to thyroidectomy
  Interventions: Procedure: Thyroidectomy

INTERVENTIONS:
Procedure: Thyroidectomy — Surgery for thyroid carcinoma

SUMMARY:
The impact of the COVID-19 pandemic has heavily influenced routine medical care. In the first months of the pandemic, healthcare authorities restricted medical care to emergency procedures, postponing elective surgical activity. Conversely, screening programmes and planned examinations have been temporarily suspended or delayed. Gradually, elective surgery and clinical activities have resumed, thanks to the weakening of the pandemic, to a better organization of the healthcare systems and to the diffusion of COVID-19 vaccines.

In the present study, we aim to evaluate the impact of the COVID-19 pandemic on surgery for thyroid carcinoma. Particularly, we aim to investigate whether the delay in operations, screening programmes, and planned examinations for patients under follow-up after thyroid surgery have led to an increased number of aggressive tumours.

To evaluate this aspect, we aim to compare the patients who had undergone thyroidectomy for thyroid cancer before the COVID-19 pandemic (from February 2019 to February 2020), during the first phase of the pandemic (from March 2020 to September 2020), and after the first phase of the COVID-19 pandemic (from October 2020 to October 2021).

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone thyroidectomy with preoperative diagnosis of thyroid cancer (cytological diagnosis, including Bethesda III, IV, IV or VI class, or high suspicion of thyroid carcinoma based on clinical and/or ultrasonographic features) during the study period (from February 2019 to October 2021)
* Patients who underwent reoperative neck surgery for local recurrence of thyroid carcinoma during the study period (from February 2019 to October 2021)

Exclusion Criteria:

* Age < 18 yo
* Incidental diagnosis of thyroid carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22974 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Incidence of aggressive thyroid cancers | 36 months
  Increase in the number of patients with aggressive thyroid carcinoma (intermediate and high risk of local recurrence, according to 2015 American Thyroid Association Guidelines on Thyroid Carcinoma), calculated as ratio between patients with aggressive thyroid carcinoma operated in pre-pandemic period and patients with aggressive thyroid carcinoma operated during covid-19 pandemic.

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Cagliari, Cagliari, CA, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Medas F, Dobrinja C, Al-Suhaimi EA, Altmeier J, Anajar S, Arikan AE, Azaryan I, Bains L, Basili G, Bolukbasi H, Bononi M, Borumandi F, Bozan MB, Brenta G, Brunaud L, Brunner M, Buemi A, Canu GL, Cappellacci F, Cartwright SB, Castells Fuste I, Cavalheiro B, Cavallaro G, Chala A, Chan SYB, Chaplin J, Cheema MS, Chiapponi C, Chiofalo MG, Chrysos E, D'Amore A, de Cillia M, De Crea C, de Manzini N, de Matos LL, De Pasquale L, Del Rio P, Demarchi MS, Dhiwakar M, Donatini G, Dora JM, D'Orazi V, Doulatram Gamgaram VK, Eismontas V, Kabiri EH, El Malki HO, Elzahaby I, Enciu O, Eskander A, Feroci F, Figueroa-Bohorquez D, Filis D, Francois G, Frias-Fernandez P, Gamboa-Dominguez A, Genc V, Giordano D, Gomez-Pedraza A, Graceffa G, Griffin J, Guerreiro SC, Gupta K, Gupta KK, Gurrado A, Hajiioannou J, Hakala T, Harahap WA, Hargitai L, Hartl D, Hellmann A, Hlozek J, Hoang VT, Iacobone M, Innaro N, Ioannidis O, Jang JHI, Xavier-Junior JC, Jovanovic M, Kaderli RM, Kakamad F, Kaliszewski K, Karamanliev M, Katoh H, Kosec A, Kovacevic B, Kowalski LP, Kralik R, Yadav SK, Kumorova A, Lampridis S, Lasithiotakis K, Leclere JC, Leong EKF, Leow MK, Lim JY, Lino-Silva LS, Liu SYW, Llorach NP, Lombardi CP, Lopez-Gomez J, Lori E, Quintanilla-Dieck L, Lucchini R, Madani A, Manatakis D, Markovic I, Materazzi G, Mazeh H, Mercante G, Meyer-Rochow GY, Mihaljevic O, Miller JA, Minuto M, Monacelli M, Mulita F, Mullineris B, Munoz-de-Nova JL, Muradas Girardi F, Nader S, Napadon T, Nastos C, Offi C, Ronen O, Oragano L, Orois A, Pan Y, Panagiotidis E, Panchangam RB, Papavramidis T, Parida PK, Paspala A, Perez OV, Petrovic S, Raffaelli M, Ramacciotti CF, Ratia Gimenez T, Rivo Vazquez A, Roh JL, Rossi L, Sanabria A, Santeerapharp A, Semenov A, Seneviratne S, Serdar A, Sheahan P, Sheppard SC, Slotcavage RL, Smaxwil C, Kim SY, Sorrenti S, Spartalis E, Sriphrapradang C, Testini M, Turk Y, Tzikos G, Vabalayte K, Vargas-Osorio K, Vazquez Renteria RS, Velazquez-Fernandez D, Vithana SMP, Yucel L, Yulian ED, Zahradnikova P, Zarogoulidis P, Ziablitskaia E, Zolotoukho A, Calo PG; THYCOVID Collaboration Group. Effect of the COVID-19 pandemic on surgery for indeterminate thyroid nodules (THYCOVID): a retrospective, international, multicentre, cross-sectional study. Lancet Diabetes Endocrinol. 2023 Jun;11(6):402-413. doi: 10.1016/S2213-8587(23)00094-3. Epub 2023 Apr 28. PMID 37127041